CLINICAL TRIAL: NCT01071057
Title: Naloxone for the Treatment of Opioid-Induced Pruritus: A Double-Blind, Prospective, Randomized, Controlled Study
Brief Title: Naloxone for the Treatment of Opioid-Induced Pruritus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mark Ansermino, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H09-03001
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pruritus
Keywords: opioid-induced pruritus; naloxone
MeSH Terms: conditions — Pruritus | interventions — Naloxone; Sodium Chloride; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naloxone/morphine (Active Comparator): Naloxone (12 µg/ml) mixed in a single infusion with morphine (1 mg/ml). The study solutions will be prepared by a pharmacist and diluted in saline to produce equal volumes to ensure proper blinding.
  Interventions: Drug: Naloxone
- saline/morphine (Placebo Comparator): Patients will be randomly assigned to one of two groups (Naloxone/morphine or saline/morphine) using computer-generated random numbers. On arrival to the PACU patients will be started on IV PCA and randomized study drug
  Interventions: Drug: Saline/Morphine

INTERVENTIONS:
Drug: Naloxone — Basal infusion of 20µg/kg/hour, bolus dose of 20µg /kg, lockout of 5 minutes with hourly maximum not to exceed 150µg /kg/hr, maximum 6 bolus doses. Subject pain relief will be assessed and documented by nursing staff and supervised by the Acute Pain Service (APS). Morphine will be titrated to subject need according to APS PCA protocol.
  Arms: Naloxone/morphine
Drug: Saline/Morphine — Basal infusion of 20µg/kg/hour, bolus dose of 20µg /kg, lockout of 5 minutes with hourly maximum not to exceed 150µg /kg/hr, maximum 6 bolus doses. Subject pain relief will be assessed and documented by nursing staff and supervised by the Acute Pain Service (APS). Morphine will be titrated to subject need according to APS PCA protocol.
  Arms: saline/morphine

SUMMARY:
The purpose of this study is to improve how we treat itching, a common side effect associated with the use of morphine pain medication. Itching is a problem experienced by up to 30% of the children treated with pain medications in the morphine family.

Despite studies demonstrating the effectiveness of using naloxone to treat itchiness in adults receiving morphine pain medications, there are not many studies in children. This study is designed to study how well naloxone works for treatment of itching in children

DETAILED DESCRIPTION:
Hypothesis: Naloxone co-administered simultaneously with standard Patient Controlled Analgesia (PCA) basal and bolus morphine will significantly reduce the incidence of Opioid Induced Pruritus (OIP) without affecting analgesia or opioid consumption in children.

Specific Objectives:

1. To determine if naloxone (12 µg/ml) mixed in a single infusion with morphine (1 mg/ml) will be effective in the prevention of opioid induced pruritus (OIP).
2. To determine if treatment with naloxone will result in attenuation of analgesia or an increase in opioid utilisation.
3. To determine if treatment with naloxone will reduce other opioid induced side effects such as nausea and vomiting.

Methods: This study is divided into two phases. Phase 1 - Although, there are studies confirming the compatibility of morphine (4 mg/mL) with naloxone (16 µg/mL) in separate infusion pumps run into the same intravenous site, there are no studies confirming the chemical and physical compatibility of morphine and naloxone in the same syringe with the standard concentrations used at BCCH. Therefore, a compatibility and stability study of naloxone and morphine solution in the same syringe will be performed.

Phase 2 - Phase 2 is a blinded clinical trial where 70 subjects will be randomized to receive either morphine mixed with naloxone or morphine mixed with placebo.With institutional review board approval, and written parental/guardian informed consent (and assent if appropriate), we will recruit children, ages 5-16 years, receiving intravenous opioids via PCA for post-operative pain control. Subjects will be evaluated every 4 hr for pain scores, frequency of vomiting, nausea, pruritus, sedation, and respiratory depression. At 24 and 48 hr, the total morphine consumption will be calculated.

Data analysis: Differences in the incidence and intensity of pruritus between the two groups will be compared. We will review side effects using the following control variables: (1) demographic data; and (2) summation of opioid use in each 4 hr period for total opioid consumption. ANOVA and crosstabs will be used where appropriate to analyze data.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-18 years of age undergoing surgery at BCCH
* ASA I - II.
* Children receiving PCA morphine.
* Informed consent/assent provided by child/parent/guardian.

Exclusion Criteria

* Children with known abnormal developmental profile.
* Children with known opioid allergy.
* Inability/failure to obtain informed consent/assent from parent/guardian/child.
* Children receiving concurrent opioids.
* Children with pre-existing pruritus from non-opioid related cause.
* Children receiving PCA hydromorphone or fentanyl.
* ASA 3 and above.
* Children who require admission to the Pediatric Intensive Care Unit (PICU). - Children involved in any investigational drug trial within the previous one month.
* Any child in the study that experiences unmanageable pruritus within the protocol time frame and is converted to hydromorphone will continue to be monitored for 48 hours. However, this will be taken into account during statistical analysis of study results. Appropriate conventional rescue medication for pruritus (diphenhydramine 0.5mg/kg IV 4hrly PRN) will be provided for any child who continues to experience pruritus.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pruritus incidence and intensity | 2 days

SECONDARY OUTCOMES:
Self-report pain scores | 2 days
Morphine, ondansetron, diphenhydramine utilization | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Lauder, Dr., Principal Investigator — University of British Columbia; Roxane Carr, Dr., Study Director — University of British Columbia; Mark Ansermino, Dr., Study Director — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Department of Anesthesia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] West N, Ansermino JM, Carr RR, Leung K, Zhou G, Lauder GR. A naloxone admixture to prevent opioid-induced pruritus in children: a randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):891-900. doi: 10.1007/s12630-015-0380-5. Epub 2015 Apr 23. PMID 25902891